CLINICAL TRIAL: NCT02785133
Title: A Polychromatic Light Emitting Diode System to Deliver Low Dose Light Directly Into a Peripheral Intravascular Catheter: A Safety and Feasibility Study
Brief Title: Safety and Feasibility of Polychromatic Light Emitting Diode for Peripheral Catheter Illumination During Peripheral Intravenous Delivery of Normal Saline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UVLrx Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVL_0001
Record Dates: First submitted 2016-01-08; First posted 2016-05-27 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Quality of Life; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Saline Solution; Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Polychromatic light emitting diode system is a non-significant risk device that administers low-dose light generated by a light emitting diode. Small adapter attaches directly to a standard 20-gauge catheter that threads a small fiber optic through the distal end of the catheter. The optic terminates at the distal end of the catheter. Polychromatic light is emitted to illuminate the catheter and site of catheter entrance. Concurrently, normal saline flows through the optic adapter and through into the 20-gauge catheter.
  Interventions: Device: UVL1000 Treatment Station; Drug: Normal Saline Solution; Device: Peripheral Catheterization

INTERVENTIONS:
Device: UVL1000 Treatment Station — Non-coherent light source administered 365 nm, 630 nm, and 530 nm at an output intensity of 0.1 mW directly into an existing intravascular 20 gauge 1.0" catheter
Drug: Normal Saline Solution — 150 ml of 0.9% Sodium Chloride Solution
Device: Peripheral Catheterization — 20-gauge 1.0" catheter

SUMMARY:
This study uses a prospective non-randomized, non-controlled design. Five-hundred (500) subjects having previously received a peripheral intravenous therapy will be enrolled into a single treatment group. The purpose of the study is to evaluate the safety, feasibility, and improved energy levels following treatment with a low-light source integrated into an existing peripheral intravascular catheter. The absence of a control group is based on the following reason:This is a pilot investigation to establish a baseline understanding of the safety, feasibility, and cursory utility of polychromatic light emitting diodes integrated into an existing 20-gauge 1.0 inch intravenous catheter to improve self-reported overall subject energy levels.

DETAILED DESCRIPTION:
This study uses a prospective non-randomized, non-controlled design. Five-hundred (500) subjects having previously received a peripheral intravenous therapy will be enrolled into a single treatment group. The purpose of the study is to evaluate the safety, feasibility, and cursory utility of a low-light source integrated into an existing peripheral intravenous catheter. The absence of a control group is based on the following reason: This is a pilot investigation to establish a baseline understanding of the safety, feasibility, and cursory utility of polychromatic light emitting diodes integrated into an existing 20-gauge 1.0 inch peripheral intravascular catheter to improve self-reported overall subject energy levels based on the change in Epworth Sleepiness scores.

Peripheral intravascular therapy has been used for decades as an effective therapy to maintain proper hydration and electrolyte levels, and has been deemed a non-significant medical procedure. Peripheral intravascular therapy can be infused with various molecular agents such as supplements (Vitamin B12) for the purpose of improving energy levels and overall quality of life. However, the use of normal saline as a standard alone helps improve hydration and cell function. Low-energy light therapy has been established as an alternative treatment for a myriad of medical conditions. Light-based therapy stimulates photoreceptors found within cells and can improve overall cellular bioenergetics. The concurrent administration of low-light therapy and peripheral intravascular normal saline therapy may serve as a viable therapy for the treatment for improvement in subject quality of life and energy levels Accordingly, this study is designed to assess the safety, feasibility, and cursory improvement in self-reported energy levels following intervention of low-light therapy integrated into a standard peripheral intravascular catheter.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form
* Ages 18-70
* Completed urine pregnancy examination with negative result
* Self-reported energy level of >4 on the Epworth sleepiness test
* No breastfeeding for 3 months prior to enrollment

Exclusion Criteria:

* Active infection along potential intravenous catheter sites
* Pacemaker
* Currently taking prescription blood thinning medications (i.e. Warfarin)
* Suffering from a chronic, progressive blood disorder, such as blood cancer (Thalassemia, Lymphoma, Myeloma, etc.)
* Use of anti-inflammatory medications on a chronic basis (i.e. ibuprofen, aspirin, and steroids)
* Suffering from blood clotting disorders (hypercoagulable condition, thrombocytosis, etc.)
* Clinically significant anxiety and/or depression
* Participated in a clinical study in the last 30 days
* Clinical Cardiac Disease
* Active Infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3063 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The use of polychromatic light therapy delivered through an intravascular catheter for the improvement in self-reported subject energy levels | Baseline and 10 weeks
  The ESS is a self-administered questionnaire with 8 questions. It provides a measure of a person's general level of daytime sleepiness, or their average sleep propensity in daily life. It has become the world standard method for making this assessment.
  The Epworth Sleepiness Scale will be used to evaluate subject energy levels at both baseline and post-procedure administration phase. Subjects will rate, on a 4-point scale (0 - 3), their usual chances of dozing off or falling asleep in 8 different situations or activities that most people engage in as part of their daily lives, although not necessarily every day. It evaluates what the chances are that they would doze off whenever they were in each situation.

SECONDARY OUTCOMES:
The improvement in subject quality of life using a five (5)-point GRA | 10 weeks
  Descriptive scale evaluating subject's perceived quality of life following treatment administration scale
Subject satisfaction based on five (5)-point satisfaction questionnaire | 10 weeks
  Self-reported overall treatment satisfaction based on perceived response from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Maloney, Study Director — Maloney Insights
Locations (1):
- Lozano Medical Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this juncture, there is no specific plan to share data with any regulatory agency for the purposes of 510k market clearance or there is no determination at this juncture to present data to the medical community (i.e. peer-reviewed publication of medical conference)